CLINICAL TRIAL: NCT05832528
Title: The Effect of a Low FODMAP Diet in Functional Dyspepsia Patients With Meal Related Symptoms on Complaint Pattern and Urinary Histamine Excretion
Brief Title: Low FODMAP Diet in FD (PDS)
Acronym: FFDU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66225
Record Dates: First submitted 2023-03-07; First posted 2023-04-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: Dietary intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FD patient (Experimental): Low-FODMAP diet in patients with FD for 6 weeks.
  Interventions: Other: Low-FODMAP diet

INTERVENTIONS:
Other: Low-FODMAP diet — 6-week Low-FODMAP diet in patients with functional dyspepsia

SUMMARY:
The goal of this dietary intervention study is to assess the efficacy and mechanisms of a low-FODMAP (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) diet in functional dyspepsia patients. The main questions it aims to answer are:

* If a low-FODMAP diet can reduce dyspeptic complaints
* How a low-FODMAP diet can reduce dyspeptic complaints in functional dyspepsia (FD).

Participants will follow a 6-week during low-FODMAP diet followed by powder reintroduction of 6 FODMAPs and 1 control substance.

DETAILED DESCRIPTION:
Functional dyspepsia Functional dyspepsia (FD) is defined as "symptoms affecting daily life which are thought to originate from the gastroduodenal region, such as postprandial fullness, early satiation, epigastric pain and burning, without underlying organic disease likely to explain the symptoms". FD is very common, with estimates of 10% to 30% prevalence in the general population, and is associated with substantial medical care costs and a considerable health economic impact. A proportion of 20%-25% of the patients with severe and refractory GI symptoms also have psychosocial co-morbidities such as anxiety, depression or somatization and severely impaired daily functioning (about 10% of these patients have work disability). This subgroup is often referred to advanced care, which may be associated with even higher health economic costs.

The pathophysiology of FD remains poorly understood and is most likely heterogeneous. The majority of FD patients have meal-related symptoms (early satiation, postprandial fullness, or epigastric pain or burning or nausea occurring or worsening after a meal). These are referred to as having Postprandial Distress Syndrome (PDS) according to the Rome IV consensus.

Leaky duodenal mucosa Duodenal and small intestinal perturbations seem to play an important role in the generation of dyspeptic symptoms. Through neuro-humoral feedback mechanisms, the duodenum plays a major role in controlling gastric functions. Mechanistic studies support the hypothesis that altered duodenal content or altered duodenal mucosal integrity are present in FD and may trigger impaired nutrient tolerance and impaired accommodation. Closely associated are signs of low grade inflammation with increased numbers of mast cells and eosinophils in the duodenal mucosa, which has been associated to symptoms of postprandial fullness and early satiation. While acute stress can increase intestinal permeability, changes in luminal factors are key candidate mechanisms to explain both mucosal permeability and immune inflammation. Duodenal acid exposure is increased in FD patients and may lead to loss of mucosal integrity and mast cell activation.

Dietary triggers The use of dietary therapeutic approaches such as the FODMAP (Fermentable Oligosaccharides, Disaccharides, Monosaccharides, And Polyols) diet to manage gastrointestinal symptoms has been frequently described and controlled studies have showed significant favorable on irritable bowel syndrome (IBS) symptoms such as abdominal pain, bloating and flatulence and it has been shown to be associated to changes in fecal microbiota. A recent study from our group showed that fructans and fructose (two of the FODMAPs) interfere with the normal meal-induced drop in intragastric pressure (IGP) and induce early postprandial occurrence of gastrointestinal symptoms, reminiscent of what happens in FD.

Measuring urinary histamine excretion McIntosh et al made an effort to identify pathophysiological mechanisms by which FODMAPs could cause gastrointestinal symptoms. They studied 20 IBS patients on a high FODMAP diet and 20 IBS patients on a low FODMAP diet. Urine samples were tested using Mass Spectrometry Analysis for metabolites that could potentially be linked to FODMAP induced post prandial distress. Patients on a low FODMAP diet had lower urinary histamine levels than IBS patients on a high FODMAP diet. The investigators hypothesize that urinary histamine excretion could be a surrogate marker for duodenal mastcell activation in patients with FD like described previously. The investigators will also measure the urinary N-methyl histamine excretion which is a more stable metabolite than histamine itself.

3. Trial objectives and Design

3.1 Trial objectives In this study, the investigators will evaluate the FODMAP diet as an alternative treatment for functional dyspepsia and explore its effect on different aspects of the pathophysiology of FD.

3.2 Primary endpoints The primary endpoint is to evaluate the efficacy of low FODMAP diet on gastrointestinal symptoms in FD.

3.3 Secondary endpoints The secondary endpoint is to explore the mechanism of action of the low FODMAP diet by evaluating duodenal mucosal permeability and urinary histamine (microgram/g creatinin in 24 hour sample) and N-methyl histamine excretion (microgram/g creatinin in 24 hour sample).

3.4 Trial Design The study design includes a 2w running up phase ('baseline'), 6 weeks of a 'strict' FODMAP diet (not blinded), followed by a 5 week 'reintroduction' phase (single blind) and, finally 2 weeks of a diet 'moderate' in FODMAP levels (not blinded). The duration of 6 weeks is based on published clinical recommendations. To support the patients' strict adherence to the diet, patients will receive a booklet with information regarding FODMAP food lists and 50 examples of FODMAP meal recipes.

The 'reintroduction' period will involve patients being challenged with 1 FODMAP group per 4 days with a wash out of 1 day after each FODMAP (4 weeks and 2 days in total). There will also be a 5 days control with glucose as a control substance. At the end of the 6 weeks of 'strict' diet, patients will receive in a blinded manner (labelled A to G) 6 containers containing the different FODMAP sugars (fructose, lactose, sorbitol, mannitol, fructans, galacto-oligosaccharides) and 1 container of glucose. The concentrations will be based on previous studies and what is commonly used in the clinical breath testing setting. These sugars can be easily dissolved in water by the patients before consumption at their homes.

Based on the patients' symptom results following each of these challenges, they will then follow the 'moderate' FODMAP diet during 2 weeks, where the FODMAPs that did not trigger any symptoms during the challenge tests can now be consumed without restriction.

24h urine, and duodenal biopsies (collected by endoscopy) will also be collected at baseline and at the end of the 6 weeks strict diet to assess alterations in duodenal integrity/inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Functional dyspepsia/ postprandial distress syndrome as per Rome IV diagnostic criteria

   * Symptom characteristics of dyspepsia (upper gastrointestinal symptoms occurring in the last 6 months and meal related (PDS))
   * Negative endoscopy (maximum 12 months old)
2. Patients must provide witnessed written informed consent prior to any study procedures being performed
3. Patients aged between 18 and 70 years inclusive
4. Male or female patients

Exclusion Criteria:

1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
2. Patients with any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years
3. Patients presenting with predominant symptoms of irritable bowel syndrome (IBS) and of gastro-oesophageal reflux disease (GERD)
4. Patients who changed their diet over the last 3 months or have previously tried the low FODMAP diet are excluded from the study.
5. Females who are pregnant or lactating are excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Effect of a low-FODMAP diet on the LPDS (Leuven-postprandial distress scale) | Measurement before and after the diet (6 weeks)
  Validated Leuven-postprandial distress scale for dyspeptic symptoms (0-15, higher scores indicating more severe symptoms)

SECONDARY OUTCOMES:
Effect of a low-FODMAP diet on urinary histamine and N-methylhistamine excretion | Measurement before and after the diet (6 weeks)
  Via 24-hour urinary collections before and after the diet, both in microgram/g creatinin in 24h urine samples
Effect of a low-FODMAP diet on duodenal mucosal integrity | Measurement before and after the diet (6 weeks)
  Measurement of TEER (trans epithelial electrical resistance) and Flux in Ussing Chambers as assessed in ussing chambers (If TEER increases then duodenal integrity increases, if flux increases then mucoal integrity decreases)
Effect of a low-FODMAP diet on duodenal low-grade inflammation | Measurement before and after the diet (6 weeks)
  Mastcell and eosinophil counting

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tack J, Talley NJ, Camilleri M, Holtmann G, Hu P, Malagelada JR, Stanghellini V. Functional gastroduodenal disorders. Gastroenterology. 2006 Apr;130(5):1466-79. doi: 10.1053/j.gastro.2005.11.059. PMID 16678560
- [Background] Lacy BE, Weiser KT, Kennedy AT, Crowell MD, Talley NJ. Functional dyspepsia: the economic impact to patients. Aliment Pharmacol Ther. 2013 Jul;38(2):170-7. doi: 10.1111/apt.12355. Epub 2013 Jun 3. PMID 23725230
- [Background] Piessevaux H, De Winter B, Louis E, Muls V, De Looze D, Pelckmans P, Deltenre M, Urbain D, Tack J. Dyspeptic symptoms in the general population: a factor and cluster analysis of symptom groupings. Neurogastroenterol Motil. 2009 Apr;21(4):378-88. doi: 10.1111/j.1365-2982.2009.01262.x. Epub 2009 Feb 12. PMID 19222761
- [Background] Talley NJ, Verlinden M, Jones M. Validity of a new quality of life scale for functional dyspepsia: a United States multicenter trial of the Nepean Dyspepsia Index. Am J Gastroenterol. 1999 Sep;94(9):2390-7. doi: 10.1111/j.1572-0241.1999.01363.x. PMID 10483997
- [Background] El-Serag HB, Talley NJ. Health-related quality of life in functional dyspepsia. Aliment Pharmacol Ther. 2003 Aug 15;18(4):387-93. doi: 10.1046/j.1365-2036.2003.01706.x. PMID 12940923
- [Background] Jones MP, Talley NJ, Eslick GD, Dubois D, Tack J. Community subgroups in dyspepsia and their association with weight loss. Am J Gastroenterol. 2008 Aug;103(8):2051-60. doi: 10.1111/j.1572-0241.2008.01935.x. PMID 18796099
- [Background] Aro P, Talley NJ, Agreus L, Johansson SE, Bolling-Sternevald E, Storskrubb T, Ronkainen J. Functional dyspepsia impairs quality of life in the adult population. Aliment Pharmacol Ther. 2011 Jun;33(11):1215-24. doi: 10.1111/j.1365-2036.2011.04640.x. Epub 2011 Mar 28. PMID 21443537
- [Background] Tack J, Piessevaux H, Coulie B, Caenepeel P, Janssens J. Role of impaired gastric accommodation to a meal in functional dyspepsia. Gastroenterology. 1998 Dec;115(6):1346-52. doi: 10.1016/s0016-5085(98)70012-5. PMID 9834261
- [Background] Carbone F, Tack J, Hoffman I. The Intragastric Pressure Measurement: A Novel Method to Assess Gastric Accommodation in Functional Dyspepsia Children. J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):918-924. doi: 10.1097/MPG.0000000000001386. PMID 27557427
- [Background] Janssen P, Verschueren S, Ly HG, Vos R, Van Oudenhove L, Tack J. Intragastric pressure during food intake: a physiological and minimally invasive method to assess gastric accommodation. Neurogastroenterol Motil. 2011 Apr;23(4):316-22, e153-4. doi: 10.1111/j.1365-2982.2011.01676.x. Epub 2011 Feb 7. PMID 21299720
- [Background] Lee KJ, Tack J. Duodenal implications in the pathophysiology of functional dyspepsia. J Neurogastroenterol Motil. 2010 Jul;16(3):251-7. doi: 10.5056/jnm.2010.16.3.251. Epub 2010 Jul 26. PMID 20680163
- [Background] Farre R, Tack J. Food and symptom generation in functional gastrointestinal disorders: physiological aspects. Am J Gastroenterol. 2013 May;108(5):698-706. doi: 10.1038/ajg.2013.24. Epub 2013 Mar 5. PMID 23458851
- [Background] Vanheel H, Vicario M, Vanuytsel T, Van Oudenhove L, Martinez C, Keita AV, Pardon N, Santos J, Soderholm JD, Tack J, Farre R. Impaired duodenal mucosal integrity and low-grade inflammation in functional dyspepsia. Gut. 2014 Feb;63(2):262-71. doi: 10.1136/gutjnl-2012-303857. Epub 2013 Mar 8. PMID 23474421
- [Background] Belic A, Grabnar I, Karba R, Mrhar A, Irman-Florjanc T, Primozic S. Interdependence of histamine and methylhistamine kinetics: modelling and simulation approach. Comput Biol Med. 1999 Nov;29(6):361-75. doi: 10.1016/s0010-4825(99)00017-7. PMID 10591171
- [Background] Walker MM, Aggarwal KR, Shim LS, Bassan M, Kalantar JS, Weltman MD, Jones M, Powell N, Talley NJ. Duodenal eosinophilia and early satiety in functional dyspepsia: confirmation of a positive association in an Australian cohort. J Gastroenterol Hepatol. 2014 Mar;29(3):474-9. doi: 10.1111/jgh.12419. PMID 24304041
- [Background] Talley NJ, Walker MM, Aro P, Ronkainen J, Storskrubb T, Hindley LA, Harmsen WS, Zinsmeister AR, Agreus L. Non-ulcer dyspepsia and duodenal eosinophilia: an adult endoscopic population-based case-control study. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1175-83. doi: 10.1016/j.cgh.2007.05.015. Epub 2007 Aug 7. PMID 17686660
- [Background] Vanuytsel T, van Wanrooy S, Vanheel H, Vanormelingen C, Verschueren S, Houben E, Salim Rasoel S, Tomicronth J, Holvoet L, Farre R, Van Oudenhove L, Boeckxstaens G, Verbeke K, Tack J. Psychological stress and corticotropin-releasing hormone increase intestinal permeability in humans by a mast cell-dependent mechanism. Gut. 2014 Aug;63(8):1293-9. doi: 10.1136/gutjnl-2013-305690. Epub 2013 Oct 23. PMID 24153250
- [Background] Raithel M, Hagel A, Albrecht H, Zopf Y, Naegel A, Baenkler HW, Buchwald F, Schultis HW, Kressel J, Hahn EG, Konturek P. Excretion of urinary histamine and N-tele methylhistamine in patients with gastrointestinal food allergy compared to non-allergic controls during an unrestricted diet and a hypoallergenic diet. BMC Gastroenterol. 2015 Apr 1;15:41. doi: 10.1186/s12876-015-0268-4. PMID 25888445
- [Background] Carbone F, Vandenberghe A, Holvoet L, Vanuytsel T, Van Oudenhove L, Jones M, Tack J. Validation of the Leuven Postprandial Distress Scale, a questionnaire for symptom assessment in the functional dyspepsia/postprandial distress syndrome. Aliment Pharmacol Ther. 2016 Nov;44(9):989-1001. doi: 10.1111/apt.13753. Epub 2016 Aug 12. PMID 27518319